CLINICAL TRIAL: NCT05707949
Title: A Multicenter, Open-label, Extension Study to Evaluate the Long-term Safety and Tolerability of Atogepant in Pediatric Subjects 6 to 17 Years of Age With Migraine
Brief Title: Long-term Extension Study to Assess Adverse Events of Oral Atogepant Tablets in Pediatric Participants (6 to 17 Years of Age) With Migraine
Acronym: Kaleidoscope
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M21-199; 2022-501099-24-00 (Other: EU CT)
Record Dates: First submitted 2023-01-24; First posted 2023-02-01 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Migraine Prophylaxis
Keywords: Migraine Prophylaxis; Atogepant; QULIPTA; AGN-241689
MeSH Terms: interventions — atogepant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atogepant Dose A (12-17 yrs) (Experimental): Participant aged 12-17 will receive oral tablets of atogepant Dose A once a day for up to 52 weeks.
  Interventions: Drug: Atogepant
- Atogepant Dose B (6-11 yrs) (Experimental): Participants aged 6-11 will receive the highest dose of oral tablets of atogepant tested in the lead-in study M21-201.
  Interventions: Drug: Atogepant

INTERVENTIONS:
Drug: Atogepant — Oral Tablet
  Other Names: QULIPTA; AGN-241689

SUMMARY:
A migraine is a moderate to severe headache on one side of the head. A migraine attack is a headache that may be accompanied by throbbing, nausea, vomiting, sensitivity to light and sound, or other symptoms. A number of treatments are available for adults with migraine but there are limited approved treatments available for participants less than 18 years of age. The main goal of the study is to evaluate the long-term safety and tolerability of atogepant in pediatric participants between the ages of 6 and 17 with migraine.

Atogepant is a medicine currently approved to treat adults with migraine (0 to 14 migraine days per month) and is being studied in pediatric participants between the ages of 6 and 17 with a history of migraine. This is a Phase 3, open-label study of atogepant in participants with a history of migraine. Participants must have completed participation in another study of atogepant (lead-in study). Participants must have 4 to 14 migraine days and less than 15 headache days for episodic migraine, and >= 15 headache days and >= 8 migraine days for chronic migraine in the 4-week screening electronic diary (eDiary; similar to a smart phone). Around 650 participants will be enrolled in the study at approximately 100 sites worldwide.

Atogepant is a tablet taken once a day by mouth. Participants between the ages of 12 and 17 will receive high dose atogepant for 52 Weeks. Participants between the ages of 6 and 11 will receive an atogepant dose determined in the lead-in study for 52 Weeks.

There may be a bigger responsibility for participants in this study. Participants will attend regular visits during the study at a hospital or clinic. The effects of treatment will be checked by medical assessments, blood tests, checking for side effects, and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between 6 and 17 years of age (inclusive), with a history of episodic (ages 6 to 17) or chronic (ages 12 to 17) migraine.
* The participant must have completed the lead-in Study M21-201, or the pharmacokinetic (PK) substudy in Study M21-201, or the lead-in Study M23-712.
* Weight is >= 20 kg (44 lbs) and < 135 kg (298 lbs).
* A history of migraine with or without aura consistent with a diagnosis according to the International Classification of Headache Disorders, 3rd Edition (ICHD-3; 2018) for at least 6 months.

Exclusion Criteria:

* Have a current diagnosis of new daily persistent headache, trigeminal autonomic cephalgia (e.g., cluster headache), or painful cranial neuropathy as defined by ICHD-3 (2018).
* Have any clinically significant hematologic, endocrine, pulmonary, renal, hepatic, gastrointestinal, cardiovascular, or neurologic disease.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 650 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2032-04 (Estimated); Study Completion 2032-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) | Up to 56 Weeks
  AE, defined as any unfavorable medical event that is temporarily related to the use of the investigational product, which does not necessarily have a causal relationship with the investigational product.
Percentage of Participants with Potentially Clinically Significant Lab Values | Up to 52 Weeks
  Percentage of participants with abnormal change in clinical laboratory test results like hematology, chemistry and urinalysis will be assessed.
Percentage of Participants with Potentially Clinically Significant Clinical 12-lead Electrocardiogram (ECG) | Up to 52 Weeks
  12-lead resting ECGs will be recorded. Parameters include heart rate, PR interval, QT interval, QRS duration, and QT interval corrected using Fridericia's formula (QTcF).
Percentage of Participants with Potentially Clinically Significant Vital Sign Parameters | Up to 52 Weeks
  Number of participants with abnormal change from baseline in vital sign measurements like systolic and diastolic blood pressure will be assessed.
Percentage of with Participants with Treatment-Emergent Suicidal Ideations with Intent, with or without a Plan (i.e., Type 4 or 5 on Columbia-Suicide Severity Rating Scale [C-SSRS]), or any Suicidal Behaviors | Up to 52 Weeks
  The C-SSRS is a clinician-rated instrument that reports the severity of both suicidal ideation and behavior. Suicidal ideation was classified on a 5-item scale: 1 (wish to be dead), 2 (nonspecific active suicidal thoughts), 3 (active suicidal ideation with any methods [not plan] without intent to act), 4 (active suicidal ideation with some intent to act, without specific plan), and 5 (active suicidal ideation with specific plan and intent). Suicidal behavior is classified on a 5-item scale: 0 (no suicidal behavior), 1 (preparatory acts or behavior), 2 (aborted attempt), 3 (interrupted attempt), and 4 (actual attempt).
Percentage of Participants with Change in Menstrual Cycle (Female Participants Only) | Up to 52 Weeks
  Female participants who have entered menarche are to be asked for the date of the first and last day of their most recent menstrual period.
Change from Baseline in Tanner Staging Score | Baseline (Week 0) through Week 52
  Tanner's staging is used to assess growth and pubertal development.
Change from Baseline in Behavior Rating Inventory of Executive Function, 2nd Edition (BRIEF 2) questionnaire | Baseline (Week 0) through Week 52
  The BRIEF 2 is an 86-item questionnaire assessing executive function. It consists of 2 indexes, Behavioral Regulation and Metacognition, which are then used to calculate an overall composite score. Higher scores indicate more executive difficulties

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (86):
- United States (35):
  - Rehabilitation & Neurological Services /ID# 250910, Huntsville, Alabama
  - Preferred Research Partners /ID# 250937, Little Rock, Arkansas
  - Advanced Research Center /ID# 251616, Anaheim, California
  - Sunwise Clinical Research /ID# 250913, Lafayette, California
  - Alliance for Research Alliance for Wellness /ID# 250911, Long Beach, California
  - Excell Research, Inc /ID# 251611, Oceanside, California
  - Lumos Clinical Research Center /ID# 251608, San Jose, California
  - Advanced Neurosciences Research, LLC /ID# 250925, Fort Collins, Colorado
  - Northwest Florida Clinical Research Group, LLC /ID# 251614, Gulf Breeze, Florida
  - Advanced Research Institute of Miami /ID# 250916, Homestead, Florida
  - My Preferred Research LLC /ID# 250931, Miami, Florida
  - Asclepes Research Centers - Spring Hill /ID# 250912, Spring Hill, Florida
  - Coastal Georgia Child Neurology /ID# 250938, Brunswick, Georgia
  - Deaconess Clinic - Gateway Health Center /ID# 250923, Newburgh, Indiana
  - College Park Family Care Center Overland Park /ID# 251609, Overland Park, Kansas
  - Michigan Headache & Neurological Institute (MHNI) /ID# 250920, Ann Arbor, Michigan
  - Proven Endpoints LLC /ID# 258083, Ridgeland, Mississippi
  - Cognitive Clinical Trials (CCT) - Papillion /ID# 251610, Papillion, Nebraska
  - Goryeb Children's Hospital /ID# 250934, Morristown, New Jersey
  - Dent Neurosciences Research Center, Inc. /ID# 250915, Amherst, New York
  - Modern Migraine MD /ID# 258082, New York, New York
  - Headache Wellness Center /ID# 251612, Greensboro, North Carolina
  - Patient Priority Clinical Sites, LLC /ID# 250922, Cincinnati, Ohio
  - CincyScience /ID# 250935, West Chester, Ohio
  - Lynn Institute of Oklahoma City /ID# 250926, Oklahoma City, Oklahoma
  - Access Clinical Trials, Inc. /ID# 250914, Nashville, Tennessee
  - FutureSearch Trials of Neurology /ID# 251613, Austin, Texas
  - 3A Research - East El Paso /ID# 250909, El Paso, Texas
  - Earle Research /ID# 250908, Friendswood, Texas
  - Family Psychiatry of The Woodlands /ID# 250936, The Woodlands, Texas
  - ClinPoint Trials /ID# 250942, Waxahachie, Texas
  - Pantheon Clinical Research /ID# 251615, Bountiful, Utah
  - Highland Clinical Research /ID# 250924, Salt Lake City, Utah
  - Office of Maria Ona /ID# 250939, Franklin, Virginia
  - Core Clinical Research /ID# 250932, Everett, Washington
- Belgium (2):
  - Uza /Id# 247885, Edegem, Antwerpen
  - AZ Sint-Jan Brugge /ID# 247527, Bruges
- Canada (2):
  - Stollery Children's Hospital /ID# 251426, Edmonton, Alberta
  - Montreal Children's Hospital /ID# 250649, Montreal, Quebec
- Denmark (3):
  - Herlev Hospital /ID# 247725, Herlev, Capital Region
  - Regionshospitalet Godstrup /ID# 247903, Herning, Central Jutland
  - Aalborg Universitetshospital /Id# 247429, Aalborg, North Denmark
- France (3):
  - CHU Amiens-Picardie Site Sud /ID# 251377, Amiens, Somme
  - Centre Hosp Intercommunal de Creteil /ID# 251199, Créteil, Val-de-Marne
  - CHU Toulouse - Hôpital des enfants /ID# 251201, Toulouse
- Hungary (2):
  - Semmelweis Egyetem /ID# 251593, Budapest, Budapest
  - Mind Klinika Kft. /ID# 251597, Budapest
- Israel (5):
  - Shamir Medical Center /ID# 256858, Beer Ya'akov, Central District
  - Hillel Yaffe Medical Center /ID# 248923, Hadera, H_efa
  - Bnai Zion Medical Center /ID# 251132, Haifa, H_efa
  - The Chaim Sheba Medical Center /ID# 248990, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 251133, Tel Aviv, Tel Aviv
- Italy (2):
  - Fondazione IRCCS Istituto Neurologico Carlo Besta /ID# 249182, Milan, Milano
  - Azienda Ospedaliera Universitaria Paolo Giaccone /ID# 249184, Palermo, Palermo
- Japan (7):
  - Konan Medical Center /ID# 254458, Kobe, Hyōgo
  - Yamaguchi Clinic /ID# 254763, Nishinomiya-shi, Hyōgo
  - Umenotsuji Clinic /ID# 254454, Kochi, Kochi
  - Sendai Headache and Neurology Clinic Medical Corporation /ID# 254212, Sendai, Miyagi
  - Tominaga Clinic /ID# 254451, Osaka, Osaka
  - Tokyo Medical University Hospital /ID# 254460, Shinjuku-ku, Tokyo
  - Tatsuoka Neurology Clinic /ID# 254456, Kyoto
- Netherlands (3):
  - Canisius-Wilhelmina Ziekenhuis /ID# 253067, Nijmegen
  - ZorgSaam Zorggroep Zeeuws-Vlaanderen /ID# 250603, Terneuzen
  - HagaZiekenhuis /ID# 251655, The Hague
- Poland (6):
  - Clinical Research Center Sp. z.o.o. Medic-R sp. k /ID# 250623, Poznan, Greater Poland Voivodeship
  - Athleticomed Sp. z o.o /ID# 250620, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Specjalistyczne Gabinety Sp. z o.o. /ID# 250625, Krakow, Lesser Poland Voivodeship
  - Indywidualna Praktyka Lekarska dr hab. med. Anna Szczepanska-Szerej /ID# 250622, Lublin, Lublin Voivodeship
  - OHA-MED sp. z o.o /ID# 250621, Warsaw, Masovian Voivodeship
  - MIGRE Polskie Centrum Leczenia Migreny Anna Gryglas-Dworak /ID# 250624, Wroclaw
- Puerto Rico (5):
  - Clinical Research Investigator Group, LLC /ID# 261251, Bayamón, Puerto Rico
  - Dr. Samuel Sanchez PSC /ID# 261670, Caguas, Puerto Rico
  - Puerto Rico Health Institute /ID# 250949, Dorado, Puerto Rico
  - Caribbean Medical Research Center /ID# 253156, San Juan, Puerto Rico
  - PRCCI Clinical Research Center /ID# 264232, San Juan, Puerto Rico
- Romania (3):
  - Spitalul Clinic de Copii Dr. Victor Gomoiu /ID# 250997, Bucharest, București
  - Spitalul Clinic de Urgenta pentru Copii Cluj Napoca /ID# 251112, Cluj-Napoca, Cluj
  - Delta Health Care S.R.L /ID# 250996, Bucharest
- Spain (4):
  - Hospital Universitario Vall d'Hebron /ID# 248457, Barcelona, Barcelona
  - Hospital Clinico San Carlos /ID# 249268, Madrid, Madrid
  - Hospital Universitario Virgen del Rocio /ID# 248633, Seville, Sevilla
  - Hospital Universitario y Politecnico La Fe /ID# 248459, Valencia, Valencia
- Sweden (2):
  - Vastra Gotealandsregionen Regionhalsan /ID# 248981, Mölnlycke
  - Sodersjukhuset /ID# 250671, Stockholm
- United Kingdom (2):
  - NHS Grampian /ID# 251474, Aberdeen
  - Stockport NHS foundation trust /ID# 261562, Stockport

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M21-199